CLINICAL TRIAL: NCT01429584
Title: Investigation Into the Effect of 0.25% Bupivacaine for Interscalene Peripheral Nerve Block vs 0.125% Bupivacaine on Pulmonary Function
Brief Title: The Effect of Interscalene Peripheral Nerve Block With 0.25% Bupivacaine vs 0.125% Bupivacaine on Lung Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Elizabeth Thackeray, Assistant Professor of Anesthesiology, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00026846
Record Dates: First submitted 2011-08-27; First posted 2011-09-07 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Diaphragm Paralysis
Keywords: bupivacaine concentration; interscalene nerve block; diaphragm function; diaphragm weakness
MeSH Terms: conditions — Respiratory Paralysis | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.25% bupivacaine (Active Comparator): interscalene nerve block with 0.25% bupivacaine
  Interventions: Drug: interscalene block with 0.125% bupivacaine
- 0.125% bupivacaine (Active Comparator): interscalene nerve block with 0.125% bupivacaine
  Interventions: Drug: interscalene nerve block with 0.25% bupivacaine

INTERVENTIONS:
Drug: interscalene nerve block with 0.25% bupivacaine — interscalene nerve block performed with 20 ml of 0.25% bupivacaine
  Arms: 0.125% bupivacaine
Drug: interscalene block with 0.125% bupivacaine — interscalene block with 20 ml of 0.125% bupivacaine
  Arms: 0.25% bupivacaine

SUMMARY:
Peripheral nerve blocks are used to provide post-operative pain relief. Nerve blocks in the neck, in the interscalene area, provide pain relief after shoulder surgery but can cause temporary weakness or paralysis of the diaphragm. The investigators hypothesized that a lower concentration of bupivacaine would cause less weakness of the diaphragm but still provide good pain relief. Lung function and pain control was studied after interscalene peripheral nerve block with 20 milliliters of 0.25% bupivacaine or 0.125% bupivacaine.

DETAILED DESCRIPTION:
Prior to placement of interscalene brachial plexus peripheral nerve block (ISPNB), diaphragm function was assessed using ultrasound as normal, no movement, or paradoxical. Room air pulse oximetry (SpO2) was recorded. Patients were randomized to receive either 0.25% bupivacaine or 0.125% bupivacaine. ISPNB was performed using a coded syringe of the study drug, so that the anesthesiologists performing the nerve block, the patient, and the nurses assessing the patient were blinded as to the concentration. Patients were given a general endotracheal anesthesia for rotator cuff repair, and opioids were administered at the discretion of the attending anesthesiologist. When patients met criteria for PACU discharge, diaphragm function was again assessed using ultrasound and room air SpO2 was recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting for outpatient rotator cuff repair
* adults
* English as the primary language

Exclusion Criteria:

* evidence of peripheral nerve damage on affected side
* refusal of peripheral nerve block
* pregnant women
* lung disease, including obstructive sleep apnea
* chronic opioid use
* mental handicap

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Thackeray, MD, MPH, Principal Investigator — University of Utah; Jeffrey Swenson, MD, Study Director — University of Utah
Locations (1):
- University of Utah Orthopaedics Center, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.25% Bupivacaine | 0.125% Bupivacaine
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.25% Bupivacaine | 0.125% Bupivacaine | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (9.3) | 53.6 (6.3) | 54.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Abnormal Lung Function
Description: Lung function was evaluated by examining diaphragm movement using ultrasound imaging and change in room air oxygen saturation (SpO2). Diaphragm movement was assessed using ultrasound as Normal (diaphragm moves caudad with inspiration), Abnormal (diaphragm does not move caudad with inspiration), and Paradoxical (diaphragm moves cephalad with inspiration). Both diaphragm function and room air SpO2 were assessed prior to any intervention to establish a baseline, and again on discharge from the PACU, within 5 hours of the completion of surgery.
Time Frame: At discharge from the post-anesthesia care unit, within 5 hours of the completion of surgery
Population: Power analysis was performed and a drop-out rate of 10% was anticipated.
Measure: Number; unit: participants w/ abnormal diaphragm fxn
Arm/Group | 0.25% Bupivacaine | 0.125% Bupivacaine
Number analyzed (Participants) | 14 | 14
participants w/ abnormal diaphragm fxn | 11 | 3

2. Secondary Outcome: Pain Relief
Description: Pain relief was assessed by recording the amount of opioid administered intraoperatively and in the PACU. The Visual Analogue Score of pain scores (0-10, with 0 being no pain and 10 being the worst pain imaginable) were recorded at the time of discharge from the PACU, within 5 hours of the completion of surgery.
Time Frame: At discharge from the post-anesthesia care unit, within 5 hours of the completion of surgery
Population: Same as other outcome measures.
Measure: Mean (Standard Deviation); unit: Visual Analogue Scale for pain
Arm/Group | 0.25% Bupivacaine | 0.125% Bupivacaine
Number analyzed (Participants) | 14 | 14
Visual Analogue Scale for pain | 0 (0) | 0.7 (1.1)

3. Secondary Outcome: Satisfaction With Pain Control
Description: A follow-up phone call was made to patients within 30 days of surgery to assess the presence of any complications related to the block and overall satisfaction with pain control. Overall satisfaction was assessed on a 7-point Likert scale of 1-not at all satisfied with pain control 2-mostly unsatisfied with pain control 3-slightly unsatisfied with pain control 4-no opinion 5-slightly satisfied with pain control 6-mostly satisfied with pain control 7-completely satisfied with pain control.
Time Frame: Within 30 days
Population: Same as other outcome measures
Measure: Mean (Standard Deviation); unit: Likert Satisfaction Scale
Arm/Group | 0.25% Bupivacaine | 0.125% Bupivacaine
Number analyzed (Participants) | 14 | 14
Likert Satisfaction Scale | 6.6 (0.5) | 6.6 (1.1)

ADVERSE EVENTS:
Arm/Group | 0.25% Bupivacaine | 0.125% Bupivacaine
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No